CLINICAL TRIAL: NCT01793194
Title: Preventing the Development of Venous Insufficiency in Pregnant Women Through Use of Compression Stockings: A Randomized Pilot Study
Brief Title: Preventing the Development of Venous Insufficiency in Pregnant Women Through Use of Compression Stockings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Sigvaris Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NA_00047720
Record Dates: First submitted 2013-02-14; First posted 2013-02-15 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Venous Insufficiency
Keywords: venous insufficiency; varicose veins; pregnancy; DVT; superficial thrombophlebitis
MeSH Terms: conditions — Venous Insufficiency; Varicose Veins | interventions — Stockings, Compression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Stocking Use (No Intervention): For pregnant women randomized to the no stocking use group, no compression stockings will be worn.
- Compression Stocking Use (Experimental): Patients who are randomized to the stocking use group (Treatment Subgroup A) will be formally measured for their stockings by a certified stocking fitter, given (at no charge) two pair of 20-30mmg Hg maternity pantyhose compression stockings, and will undergo a brief tutorial regarding how to put the stockings on. Each patient will be instructed to wear the stockings on a daily basis, during the day.
  Interventions: Other: Compression Stockings

INTERVENTIONS:
Other: Compression Stockings — 20-30mmg Hg maternity pantyhose compression stockings
  Arms: Compression Stocking Use

SUMMARY:
Problem: Approximately 4 million live births occur in the United States each year. Pregnancy causes many physical changes in the mother, including venous distension, increased ability to form blood clots, and hormonal changes. Data suggest that these factors help cause venous insufficiency (when the veins do not adequately return blood from the extremities to the torso). As venous insufficiency progresses, complications follow, the most severe of which include superficial thrombophlebitis and deep venous thrombosis (DVT, or blood clots). Although the fear of DVT has been well publicized, its prevention and prevalence in pregnant women has not been well-studied.

The exact cause of venous insufficiency is not known. However, known risk factors include being female and hormonal changes associated with oral contraceptive use, certain hormone replacement medications, and pregnancy. Being pregnant places the mother at additional risk for developing venous insufficiency.

Compression stockings are used to manage the condition, but this is by no means standard of care despite their easy use and safety. The medical community's understanding of how compression stockings work is largely theoretical; however, it is believed that the compression works by preventing venous hypertension in the lower legs, thereby preventing venous insufficiency and its associated complications.

Research hypothesis: The investigators hypothesize that compression stocking use will be associated with lower incidence of varicose veins and, in those patients who already have varicose veins, lower incidence of complications associated with venous insufficiency. Further, the investigators believe that compression stocking use will be associated with a lower incidence or lessening of symptoms associated with venous insufficiency.

Importance: An undetected DVT can be fatal. Even if detected promptly, DVT is associated with long term health problems. Treatment of a DVT requires anticoagulation which can be risky to both mother and fetus. The prevention or reduction of DVT in pregnant women through use of compression stockings would revolutionize their care. Further, this intervention is safe and noninvasive.

The investigators propose to conduct a randomized, pilot study comparing pregnant women without and with varicose veins randomized to wear compression stockings to a similar group of participants randomized to no compression stocking use.

DETAILED DESCRIPTION:
Problem: There are approximately four million live births in the United States annually. Pregnancy induces multisystemic physiologic changes in the mother as her body accommodates the growing fetus. Known physiologic alterations include venous distension, hypercoagulability, and hormonal changes. Anecdotal data suggests that these particular factors precipitate the development of venous insufficiency. As venous insufficiency progresses, complications ensue, the most severe of which include superficial thrombophlebitis and deep venous thrombosis. Although the fear of deep venous thrombus (DVT) has been well publicized, its prevention and actual prevalence in the pregnant population has not been adequately studied.

The precise mechanism of venous insufficiency has yet to be elucidated. However, several known risk factors exist. They include female gender and hormonal changes associated with elevated progesterone levels such as oral contraceptive use, certain exogenous hormonal replacement medications, and pregnancy. Clearly, the pregnant state places the mother at additive risk for subsequent development of venous insufficiency.

Medical management of venous insufficiency consists of compression stocking use, and some physicians do recommend their use to pregnant patients. However, this practice is by no means standard of care, despite its noninvasive application and safety. The precise mechanism through which compression stockings work is largely theoretical; however, it is believed that the extrinsic graduated compression works by preventing venous hypertension in the distal lower extremity, thereby preventing venous insufficiency and its associated complications.

Research hypothesis: The investigators hypothesize that compression stocking use will be associated with lower incidence of varicose veins and, in those patients who already have varicose veins, lower incidence of complications associated with venous insufficiency, particularly superficial thrombophlebitis and deep venous thrombosis (DVT). Further, the investigators believe that compression stocking use will be associated with a lower incidence or lessening of symptoms associated with venous insufficiency, such as edema, fatigue, venous stasis dermatitis, and venous neuropathy (burning).

Importance: While some may feel that varicose veins, edema, fatigue, and other outcomes are unimportant, an undetected DVT is commonly a fatal event. Even if detected promptly, DVT is associated with long term morbidity, such as post thrombotic syndrome which can occur in up to 30% of those patients diagnosed with a DVT. Treatment of a DVT requires anticoagulation which, although essential, carries significant risk to both mother and fetus. The prevention or reduction in incidence of DVT in this population merely with compression stocking use would revolutionize care in the pregnant population. Further, this intervention is safe and noninvasive.

The investigators propose to conduct a randomized, pilot study comparing pregnant women without (Group 1) and with (Group 2) varicose veins randomized to wear compression stockings (Treatment Subgroup A) to a similar group of participants randomized to no compression stocking use (Control Subgroup B).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women 18-45 years of age.
* Fetal gestation between 8-20 weeks.
* Patient is seeking care for the pregnancy at one of the study locations (Johns Hopkins East Baltimore Campus, Johns Hopkins Bayview Medical Center, and Johns Hopkins at White Marsh).
* Ability to complete informed consent and willingness to comply with protocol (return for all follow-up visits & participate in phone interviews).

Exclusion Criteria:

* Inability to wear compression stockings.
* Women who currently have been prescribed to wear compression stockings by a medical professional.
* Chronic dermatological condition (i.e. psoriasis).
* Chronic deep vein thrombus or chronic phlebitis.
* In women with varicose veins: Presence of primary outcome (superficial thrombophlebitis or DVT) on first visit ultrasound.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2014-08-24 (Actual); Study Completion 2014-08-24 (Actual)

PRIMARY OUTCOMES:
Incidence of varicose veins | 8 weeks post-partum
  In pregnant women who do not have varicose veins (Group 1): To quantify and compare the incidence of varicose veins between participants randomized to the compression stocking use group (Group 1A) and those randomized to the no compression stocking use group (Group 1B).
Incidence of superficial thrombophlebitis and DVT | 8 weeks post-partum
  In pregnant women who already have varicose veins (Group 2): To quantify and compare the incidence of superficial thrombophlebitis and DVT between those randomized to the compression stocking use group (Group 2A) and those randomized to the no compression stocking use group (Group 2B).

SECONDARY OUTCOMES:
Incidence of symptoms of venous insufficiency | 8 weeks post-partum
  For All Groups: To quantify and compare the incidence of symptoms of venous insufficiency in pregnant women between the treatment and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Heller, MD, Principal Investigator — Div. of Vascular Surgery, Johns Hopkins University School of Medicine
Locations (1):
- Johns Hopkins Bayview Medical Center and Johns Hopkins Hospital, Baltimore, Maryland, United States